CLINICAL TRIAL: NCT04479046
Title: Evaluating the Efficiency of Newly Designed Prefabricated PMMA Crowns for Restoring Primary Teeth in Comparison to Stainless Steel and Zirconia Crowns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nada Aboushady, Assistant Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAP202
Record Dates: First submitted 2019-12-27; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Decay, Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stainless steel crowns (Active Comparator): 3M ESPE
  Interventions: Other: PMMA crowns
- Zirconia crowns (Experimental): Nu Smile
  Interventions: Other: PMMA crowns
- PMMA crowns (Experimental): Dental Direkt
  Interventions: Other: PMMA crowns

INTERVENTIONS:
Other: PMMA crowns — New type of pediatric crowns

SUMMARY:
Evaluation of PMMA pediatric crowns

DETAILED DESCRIPTION:
The aim of the present study is to evaluate the PMMA crowns regarding the following aspects:

I. Clinical evaluation of PMMA crowns regarding wear of opposing teeth when compared to zirconia crowns and stainless steel crowns after 6 months, and 12 months.

II. Color stability of PMMA crowns and zirconia crowns after 6 months, and 12 months.

III. Gingival health of restored teeth after 6 months, and 12 months. IV. Patient's satisfaction regarding the appearance and clinical performance of PMMA crowns when compared to stainless steel crowns and zirconia crowns through a given questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Children included in the study should conform to the following criteria:

  1. Aged 5-8 years old
  2. Medically free
  3. Patient should suffer from extensively decayed primary lower second molar that will undergo pulpotomy.
  4. The anticipated exfoliation date of the selected primary teeth has to be more than 12 months from the date of the study start.

     Exclusion Criteria:

     Children with the following criteria will be totally excluded from the study:

  <!-- -->

  1. Children who are extremely uncooperative and difficult to manage.
  2. Children suffering from any medical conditions that can't be managed in the clinic.
  3. Teeth with decay extending beneath the free gingival margin.
  4. Teeth that were grossly broken down, that cannot be restored.
  5. Presence of uncontrolled bleeding.
  6. Clinical or radiographic evidence of non-vitality such as presence of an abscess or a sinus, obvious discoloration, and premature hypermobility.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Gingival health | 6 months
  Plaque index
Crown survival | 6 months
  Fracture

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Ain Shams University, Heliopolis, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided